CLINICAL TRIAL: NCT00079807
Title: Painful HIV Neuropathy: Treatment With Alpha-Lipoic Acid
Brief Title: Painful HIV Neuropathy and Alpha-Lipoic Acid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001775 (NIH); MannJ
Record Dates: First submitted 2004-03-15; First posted 2004-03-16 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: HIV; Peripheral Neuropathy
Keywords: HIV; Peripheral neuropathy; Alpha-Lipoic Acid; ALA; Complementary Therapies
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Thioctic Acid

INTERVENTIONS:
Drug: Alpha-Lipoic Acid

SUMMARY:
HIV is associated with painful peripheral neuropathy. Disability is often significant. Alpha-Lipoic Acid's antioxidant properties may have benefit in this condition.

DETAILED DESCRIPTION:
HIV is associated with painful distal peripheral polyneuropathy in up to 35-50% of those without AIDS and in more than 70% of those with advanced disease. The condition is progressive but may be halted with disease remission. Disability is often significant. Peripheral nerve axons and sensory neuron cell bodies in the dorsal root ganglia are the principal targets of the process leading to symptoms. Alpha-lipoic acid occurs naturally in every cell of the body. In high concentrations it acts as an anti-oxidant which regenerates other anti-oxidants and promotes glutathione synthesis. Clinical studies for diabetic neuropathy have shown significant benefit at daily oral doses that are well-tolerated.

This placebo-controlled study is designed to evaluate the effects of daily oral alpha-lipoic acid supplements (600mg, three times per/day) plus standard medical care in the treatment of painful HIV-associated neuropathy over a 24-week period in adult subjects. Possible benefits of the study include reduction in pain and disability, reduced use of medications, and enhanced cellular metabolism.

ELIGIBILITY:
Inclusion Criteria:

* HIV-seropositive
* Distal peripheral sensory neuropathy as diagnosed by a neurologist with pain or paresthesia, with or without numbness or weakness
* Able to understand and participate in protocol activities
* Able to give informed consent
* Under the care of a UNC ID Clinical physician for at least 2 months
* Able to document pain characteristics, use of pain medications, and other assessment instruments and characteristics
* On stable antiretroviral therapy (or none) for 12 weeks prior to enrollment
* No changes in peripheral neuropathy pharmacologic treatment for 12 weeks prior to enrollment

Exclusion Criteria:

* Any significant cognitive impairment or psychosis
* Pregnancy or anticipated pregnancy (women of child-bearing potential must agree to use birth control for the duration of the study)
* Undergoing any current treatment for malignancy, including chemotherapy or radiation therapy within the past year
* Concurrent or prior use of a-LA
* Known non-HIV risk factors for peripheral neuropathy, such as DM, B12/folate deficiency; thyroid dysfunction; hx of exposure to lead, mercury, arsenic, thallium (prior diagnostic tests permitted), other heavy metals or complex hydrocarbons
* Use of metronidazole, isoniazid or other furantoins
* Suspected or documented thiamin deficiency
* Active alcoholism
* Allergy to a-LA
* Hx of 'significant' use of anti-oxidant supplements during the two months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mann, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States